CLINICAL TRIAL: NCT06424054
Title: Mitigating Toxicity of (Neo)Adjuvant Chemotherapy by Applying Electronic Health Portal-mediated Interactive Monitoring of Patient-reported Side Effects: the Prospective Randomized eChemoCoach Trial
Brief Title: Mitigating Toxicity by Electronic Health Portal-mediated Interactive Monitoring of Patient-reported Side Effects
Acronym: eChemoCoach
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Noordwest Ziekenhuisgroep (Other)
Collaborators: Comprehensive Cancer Centre The Netherlands (Other); University of Twente (Other); Dutch Cancer Society (Other); Borstkanker Onderzoek Groep (Network)
Responsible Party: Principal Investigator, Mathijs Hendriks, MD, Principal investigator, Noordwest Ziekenhuisgroep
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-01/15741 (KWF-grant)
Record Dates: First submitted 2024-04-09; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; eHealth; Symptom Monitoring; Self Management
Keywords: Breast Cancer; remote monitoring; emonitoring; eHealth; symptom management; symptom monitoring
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: A clinical randomized controlled trial will be performed in 746 breast cancer patients treated with (neo-)adjuvant chemotherapy. Patients will be randomized to the intervention group, using the eChemoCoach in addition to standard of care monitoring to manage side effects or are randomized to solely standard of care monitoring.
Masking Description: This is a open label study since blinding is not possible as healthcare professionals will receive the CTC gradation based on the reported side effects in the intervention group and are obligated to act on these reports.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eChemoCoach Group (Experimental): Patients assigned to the intervention arm fill in the eChemoCoach questionnaires. They will be asked to report their side effects at baseline (2 - 4 days before their first chemotherapy cycle) and weekly thereafter. Moreover, they can report their symptoms at any time in case of potential toxicity, with a maximum of once a day. Non-responders receive reminders. Both intervention and control groups receive standard monitoring and coaching, including pre-scheduled checks for side effects before chemotherapy. Patients in both groups are asked to complete questionnaires measuring the impact on HRQoL, anxiety, distress, and patient empowerment at baseline, 10 weeks, and 20 weeks post-chemotherapy initiation. Usability of the eChemoCoach will be assessed through an online survey for patients and healthcare professionals using the System Usability Scale
  Interventions: Other: eChemoCoach
- Control group (No Intervention): Patients in the control group receive standard of care. Both intervention and control groups receive standard monitoring and coaching, including pre-scheduled checks for side effects before chemotherapy. Patients in both groups are asked to complete questionnaires measuring the impact on HRQoL, anxiety, distress, and patient empowerment at baseline, 10 weeks, and 20 weeks post-chemotherapy initiation.

INTERVENTIONS:
Other: eChemoCoach — the eChemoCoach is an electronic questionnaire which is accessible for patients via the secured electronic health portal (EHP) of the EHR, which is CE-certified. By utilizing the eChemoCoach, patients (for this project we focus on breast cancer patients) have the ability to complete a questionnaire on a daily basis, when experiencing side effects. The eChemoCoach has the potential to evaluate the severity of adverse effects based on the CTCAE criteria and triage them, mimicking the decision-making process of a HCP through computer adaptive testing (CAT). Upon completing the questionnaire, the eChemoCoach translates the responses for each specific side effect into corresponding CTCAE grades. The tool then promptly offers patients personalized advice, tailored to their individual condition.
  Arms: eChemoCoach Group

SUMMARY:
Chemotherapy induces side effects varying in severity, impacting patients' quality of life and necessitating unplanned hospital care. Patient-reported outcomes (PROs) could aid in early detection and management of side effects. However, existing PRO monitoring lacks triage capabilities, leading to clinician involvement and suboptimal symptom management. The investigators propose eChemoCoach, an electronic questionnaire integrated into the electronic health portal, offering real-time symptom assessment and personalized advice based on CTCAE criteria. Our study aims to assess the impact of eChemoCoach on non-hematological CTCAE ≥ 3 graded side effects in early breast cancer patients undergoing chemotherapy. This is a randomized controlled trial involving 746 patients that will evaluate the eChemoCoach's efficacy compared to standard monitoring. Phase one will validate questionnaires and assess usability, while phase two focuses on the primary outcome. Te investigators anticipate reduced severe side effects, thereby enhancing patients' quality of life, reducing stress, and minimizing hospital visits.

DETAILED DESCRIPTION:
Problem description: The aim of (neo)adjuvant chemotherapy is to increase survival. Therefore, treatment adherence is important. However, patients may experience treatment-related side-effects. In current practice, clinicians evaluate toxicity just a few days before the next chemotherapy is scheduled. Monitoring and timely anticipation of chemotherapy related side-effects may prevent escalation of toxicity, increase treatment adherence and reduce the decline in quality of life. Evaluating toxicity more frequently and on-demand could be a solution to reduce severe toxicity. Therefore, patients should receive a direct advice when experiencing side-effects. However, without interference of a health care professional, this is not possible in standard care.

Solution / research direction: There is increasing evidence that incorporating patient reported outcomes (PROs) in clinical care enhances symptom monitoring in cancer patients. Therefore, it is desirable to develop and investigate an electronic smart-phrased side-effects questionnaire which: 1) delivers a real-time personalized advice to the patient, based on CTCAE grading, after the questionnaire is completed and 2) is accessible for patients using an electronic health portal (EHP) of the electronic health record (EHR) to integrate the PRO data into the EHR.

Aim / hypothesis: To investigate the effect of adding weekly EHP-mediated monitoring of chemotherapy related side-effects based on CTCAE grading using smart-phrased electronic PRO side-effects questionnaires to standard of care monitoring of side-effects, on the occurrence of CTCAE >= grade 3 toxicity.

Plan of investigation: To conduct a pilot study to validate the smart-phrased ePRO side-effects questionnaire. Thereafter, a multicenter clinical randomized trial will start where patients with breast cancer qualifying for (neo)adjuvant chemo(immune)therapy will be randomized to real-time EHP-mediated monitoring of side-effects using a novel smart-phrased ePRO side-effects questionnaire in addition to standard of care monitoring, or to standard of care monitoring solely. Primary objective is the overall rate of CTC grade >=3 non hematological toxicity between both arms. Secondary objectives include relative dose intensity, health-related quality of life, experienced distress, the number of unplanned health care usage and costs.

Expected outcome: The investigators hypothesize that adding weekly EHP-mediated monitoring of side-effects using ePRO side-effects questionnaires will significantly lower the occurrence rate of CTCAE grade >=3 non-hematological toxicities.

ELIGIBILITY:
Inclusion Criteria:

* - Starting (neo)adjuvant treatment with chemotherapy for breast cancer according to one of the below mentioned treatment protocols:

  * Four cycles of doxorubicin 60mg/m2 and cyclophosphamide 600mg/m2 (AC) dose dense q 2 weeks, followed by twelve cycles of weekly paclitaxel 80mg/m2 (also in combination with carboplatin AUC6 q 3 weeks)
  * Nine cycles q 3 weeks of paclitaxel 80mg/m2 on day 1 and 8, carboplatin AUC 3 on day 1 and 8, trastuzumab 8mg/kg loading dose (followed by doses of 6mg/m2 at subsequent cycles) on day1 and pertuzumab loading dose of 840mg (followed by doses of 420mg at subsequent cycles) on day 1
* Age ≥ 18 years
* WHO PS ≤1
* Capable of using the EHP or get help in case of low (e-)health literacy. This includes being capable of login using DigiD, a system used by the Dutch government to verify the identity of a person
* Being able to read or get help from a relative in case of illiteracy

Exclusion Criteria:

* - Participation in a trial with an investigational product (because more frequent and structured symptom reporting is performed in these studies).
* Patients who have been treated with chemotherapy in the past (since these patients are at higher risk for developing side effects of current chemotherapy).
* Patients that already started with their chemotherapy cycle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
The occurrence of any non-hematological side effects grade ≥3 | Up to 30 weeks after start chemotherapy
  The occurrence of any non-hematological side effects grade ≥3 during neo-adjuvant or adjuvant treatment

SECONDARY OUTCOMES:
Toxicity patterns | Up to 30 weeks after start chemotherapy
  Time to occurrence of both grade 2 and grade ≥3 toxicity will be analyzed with a Kaplan-Meier curves.
  Occurrence of grade 2 side effects during (neo)adjuvant will be presented as numbers with percentages for patients in both study groups.
Relative dose intensity (RDI) | Up to 30 weeks after start chemotherapy
  For analyzing the RDI, the RDI will be calculated for each chemotherapeutic agent and presented as mean with standard deviations (SD) (for a description of calculation of the RDI see the objective section paragraph 2.0). The RDI will be calculated per cycle. The RDI will be compared between the intervention and the control group.
HRQOL | on baseline, 10 and 20 weeks after start of chemotherapy
  Health-related quality of life measured by the Quality of Life Questionnaire (QLQ-C30s). Scale is ranging from 1 to 4. 1 = not at all, 4 = very much. Higher scores mean a worse QOL.
Patient experienced anxiety | on baseline, 10 and 20 weeks after start of chemotherapy
  Patient experienced anxiety measured using the Hospital Anxiety and Depression Scale. Scale is ranging from 0 to 3. 0 = often, 3 = never. Higher scores means a less worse Hads score.
Patient empowerment | on baseline, 10 and 20 weeks after start of chemotherapy
  Patient empowerment using Patient Activation Measure (PAM13) questionnaire. Ranging from 0 to 3. 0 = I do not agree, 3= I totally agree. A lower score is worse.
Patient experienced stress | on baseline, 10 and 20 weeks after start of chemotherapy
  Patient experienced stress using a distress thermometer. Ranging from 0 to 10 per problem. 0 = no problem, 10 = worst. A higher score means more stress.
Unplanned Care | Up to 30 weeks after start chemotherapy
  The amount of unplanned hospital care will be presented as median (IQR) and will be analyzed by comparing the number of admissions, unplanned visits, days of hospital admissions between the intervention and control group using Poisson regression analysis.
Validation of eChemoCoach questionnaires | During the first year of the study
  Cognitive interviews will be analyzed with thematic content analysis. Agreement between professional triage estimations and eChemoCoach will be quantified using Cohen's Kappa coefficient. A semi qualitative assessment will be conducted, comparing the patient-reported adverse effects using eChemoCoach with medical professionals' CTCAE severity assessments. Interviews will be analyzed with thematic content analysis.
Usability | After inclusion of all intervention patients
  The System Usability Scale will be used for global assessment of the eChemoCoach. usability. Usability will also be assessed by healthcare professionals from participating. sites. The SUS is a 10 item questionnaire with 5 response options. Ranging from strongly disagree to strongly agree. The average SUS score from all 500 studies is a 68. A SUS score above a 68 would be considered above average and anything below 68 is below average.
Agreement eChemoCoach-reported grades and those reported by PRO-CTCAE, HCPs, and the Dutch translation of CTCAE | Up to 30 weeks after start chemotherapy
  To assess the concordance among eChemoCoach-reported grades, PRO-CTCAE, and CTCAEs graded by healthcare professionals (HCPs), we employ the eChemoCoach platform for patient experienced symptom data collection. Each questionnaire administered includes the eChemoCoach and the PRO-CTCAE questionnaire, facilitating immediate and direct comparison of both outcomes. HCPs will document symptom grading in patient files using standardized CTCAE forms. HCPs will grade the severity on pre-planned checks (standard of care) and when necessary in case of severe side effects.

IPD SHARING:
Plan to Share IPD: Yes